CLINICAL TRIAL: NCT03192839
Title: Early DHA Supplementation in Very Low Birth Weight Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mead Johnson Nutrition (Industry)
Collaborators: North Shore Research Institue (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 6039
Record Dates: First submitted 2017-06-19; First posted 2017-06-20 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Prematurity
MeSH Terms: conditions — Premature Birth | interventions — Fatty Acids, Unsaturated

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low dose PUFA (Experimental)
  Interventions: Other: Low dose PUFA
- High dose PUFA (Experimental)
  Interventions: Other: High dose PUFA
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Low dose PUFA — Low dose PUFA
  Arms: Low dose PUFA
Other: High dose PUFA — High dose PUFA
  Arms: High dose PUFA
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This clinical trial will evaluate the effects of giving supplements of PUFA to premature infants.

ELIGIBILITY:
Inclusion Criteria:

* Very low birth weight infants weighing less than 1500 grams
* Consent signed within 72 hours of life

Exclusion Criteria:

* Infants with know metabolic disorder
* Infants with known congenital GI anomaly
* Infants who are deemed to be inappropriate for enrollment per attending neonatologist

Max Age: 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-07-09 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Red Blood Cell polyunsaturated fatty acids (PUFA) levels | 2 weeks of age

SECONDARY OUTCOMES:
Red Blood Cell PUFA levels | 8 weeks of age
Feeding tolerance | 8 weeks
  Full enteral feed of 120 kcal/kg/day
Incidence of necrotizing enterocolitis | 8 weeks
Incidence of bronchopulmonary dysplasia | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Cooper, M.D, Study Director — Mead Johnson Nutrition
Locations (2):
- United States (2):
  - Rush University Medical Center, Chicago, Illinois
  - North Shore University Health System, Evanston, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Frost BL, Patel AL, Robinson DT, Berseth CL, Cooper T, Caplan M. Randomized Controlled Trial of Early Docosahexaenoic Acid and Arachidonic Acid Enteral Supplementation in Very Low Birth Weight Infants. J Pediatr. 2021 May;232:23-30.e1. doi: 10.1016/j.jpeds.2020.12.037. Epub 2021 Feb 20. PMID 33358843